CLINICAL TRIAL: NCT03409471
Title: Human Papillomavirus(HPV) Test of Urine and Self Collected Vaginal Samples for Cervical Cancer Screening Study
Brief Title: HPV Test of Urine and Self Collected Vaginal Samples for Cervical Cancer Screening Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Cheil General Hospital and Women's Healthcare Center (Other); Samsung Medical Center (Other); Korea University (Other)
Responsible Party: Principal Investigator, Jae Kwan Lee, Professor, Korea University Guro Hospital
Other Study IDs: K2017-9243 (HPV Ur SELF)
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: ASC-US; LSIL
Keywords: Urine; Cervical Intraepithelial Neoplasia; Self-Sampling; HPV Testing; Cervical Cancer Screening; ASCUS; LSIL
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine sample, vaginal self-sample and cervical cell sample collected by a gynecologist. No human DNA is extracted from the samples but the samples can contain HPV DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Flocked Swab — At the colposcopy clinic, vaginal self-sample will be collected with the Flocked Swab (Noble Bioscience, Inc., Korea).
Device: Cervical Brush — Physician collected cervical sample will be collected also at the colposcopy center with the Cervical Brush (Noble Bioscience, Inc., Korea).
Diagnostic Test: HPV assay — The hrHPV assay used, will be the Roche Cobas® 4800 HPV test, Anyplex™ II HPV HR detection kit and Realtime HPV HR-S Detection kit.

SUMMARY:
This study is a prospective observational study of human papillomavirus (HPV) testing using urine and self-collected vaginal samples for women who have atypical squamous cells of undetermined significance(ASCUS) or low grade squamous intraepithelial lesion(LSIL) on Pap test. Among women who are diagnosed with ASCUS and LSIL, HPV test is performed by collecting urine and self-collected vaginal sample in standardized condition before colposcopy, and evaluation will be performed as a primary screening test with cytology triage.

DETAILED DESCRIPTION:
The samples are collected from patients referred to colposcopy because of prior cervical abnormalities on Pap test such as ASCUS and LSIL. The patient takes at home urine samples on the morning of visit to the colposcopy center. At the colposcopy center, self-collected vaginal samples are taken by the patient herself with a plastic brush (Flocked Swab, manufactured by Noble Bioscience, Inc.). Finally, the gynecologist takes a cervical sample with a plastic brush (Cervical Brush, manufactured by Noble Bioscience, Inc.).

Physician collected cervical samples, self-collected vaginal samples and urine samples are used to perform HPV testing with Roche Cobas® 4800 HPV test, Anyplex™ II HPV HR detection kit and Realtime HPV HR-S Detection kit.

The Anyplex™ II HPV HR detection kit (manufactured by Seegene. Inc, Korea) is a new, multiplex, real-time polymerase chain reaction assay to detect individual 14 high-risk. (HR) human papillomavirus (HPV) types in a single tube.

The Roche Cobas® 4800 HPV test (manufactured by Cobas) is a novel molecular method based on real-time PCR (RT-PCR), with a fully automated system allowing quick and efficient sample processing. Cobas can detect the human papillomavirus type 16(HPV16), the human papillomavirus type 18(HPV18), 12 other high-risk HPVs (hrHPVs) (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, and -68, as a pooled result), and the β-globin control independently in the same PCR.

Realtime HPV HR-S Detection kit (manufactured by Sejong Biomed Co, Korea) is a new, real-time polymerase chain reaction assay to detect HPV 16, HPV 18, 12 other high-risk HPVs (HPV31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66, and -68). Real-time HPV HR-S Detection Kit is based on accurate real-time PCR method as described, and it can detect 14 kinds of HPV type detection in a single test (HPV 16/18 genotype and others (UDG) -dUTP) system for the prevention of contamination, and a control agent (hemoglobin DNA, a human-derived DNA) as a whole process control was introduced into a high-risk genotype (12 genotypes other than HPV 16/18). It has high sensitivity and specificity for detection of high risk genotypes by increasing the reliability of the results.

The main goal of this study is to determine whether HPV testing using urine and self-collected sample is sensitive to detecting precancerous lesions such as cervical intraepithelial neoplasia(CIN)2/3 in patients diagnosed with ASCUS and LSIL on the Pap test. The colposcopy and histological findings will be used as the gold standard. In addition, the relative sensitivity and specificity for detecting HPV16, HPV18 and high risk HPV will be determined for each of the three HPV tests using urine and self-collected samples compared with the HPV tests using physician-collected samples.

ELIGIBILITY:
Inclusion Criteria:

* Women with previous abnormal Pap test results (ASCUS, LSIL)
* Women between the ages of 20 and 60

Exclusion Criteria:

* Hysterectomised women
* Women with known pregnancy
* Non-consenting women
* Women that are not able to understand and to sign the informed consent
* Women who diagnosed and treated for cervical cancer or other malignancies
* Concurrent diseases that are immunosuppressed or require the use of immune-suppressants

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 300 women visited to a participating colposcopy centers (Korea University Guro Hospital, Korea University Ansan Hospital, Seoul Samsung Medical Center and Cheil General Hospital and Women's Healthcare Center), because of a previous abnormal Pap test result (ASCUS, LSIL), will be enrolled after obtaining informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical accuracy | Within 6 months after study completion
  Absolute sensitivity and specificity for finding underlying cervical intraepithelial neoplasia(CIN)2+ of HPV testing(Roche Cobas® 4800 HPV test, Anyplex™ II HPV HR detection kit and Realtime HPV HR-S Detection kit) on urine, self- and clinician-collected samples.

SECONDARY OUTCOMES:
Clinical accuracy | Within 6 months after study completion
  Relative sensitivity and specificity of hrHPV testing on vaginal self-samples and urine sample vs clinician-collected samples.
Analytical performance | Within 6 months after study completion
  Concordance of the presence of HPV16, 18 and other high risk HPV genotyping results applied on urine, self- and clinician-collected samples

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kwan Lee, MD, Ph.D., Principal Investigator — Professor
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung S, Lee B, Lee KN, Kim Y, Oh EJ. Clinical Validation of Anyplex II HPV HR Detection Test for Cervical Cancer Screening in Korea. Arch Pathol Lab Med. 2016 Mar;140(3):276-80. doi: 10.5858/arpa.2015-0117-OA. PMID 26927723
- [Background] Cui M, Chan N, Liu M, Thai K, Malaczynska J, Singh I, Zhang D, Ye F. Clinical performance of Roche Cobas 4800 HPV Test. J Clin Microbiol. 2014 Jun;52(6):2210-1. doi: 10.1128/JCM.00883-14. Epub 2014 Apr 9. PMID 24719443
- [Background] Stanczuk GA, Currie H, Baxter G, Foster A, Gibson L, Graham C, Cuschieri K. Cobas 4800 HPV detection in the cervical, vaginal and urine samples of women with high-grade CIN before and after treatment. J Clin Pathol. 2015 Jul;68(7):567-70. doi: 10.1136/jclinpath-2014-202851. Epub 2015 Apr 15. PMID 25878328
- [Background] Connor RJ. Sample size for testing differences in proportions for the paired-sample design. Biometrics. 1987 Mar;43(1):207-11. PMID 3567305
- [Background] Stanczuk G, Baxter G, Currie H, Lawrence J, Cuschieri K, Wilson A, Arbyn M. Clinical validation of hrHPV testing on vaginal and urine self-samples in primary cervical screening (cross-sectional results from the Papillomavirus Dumfries and Galloway-PaVDaG study). BMJ Open. 2016 Apr 25;6(4):e010660. doi: 10.1136/bmjopen-2015-010660. PMID 27113237
- [Background] Guan P, Howell-Jones R, Li N, Bruni L, de Sanjose S, Franceschi S, Clifford GM. Human papillomavirus types in 115,789 HPV-positive women: a meta-analysis from cervical infection to cancer. Int J Cancer. 2012 Nov 15;131(10):2349-59. doi: 10.1002/ijc.27485. Epub 2012 Mar 20. PMID 22323075
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571